CLINICAL TRIAL: NCT02766231
Title: A Multicentre, Prospective Study Evaluating Clinical, Radiographic and Patient-reported Outcomes of Total Knee Arthroplasty With Physica CR or Physica PS Prosthesis
Brief Title: Physica CR and Physica PS Clinical Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: K-09
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Physica CR: Patients who have undamaged and functional collateral and posterior cruciate ligaments for the group requiring Physica CR
  Interventions: Device: Physica CR
- Physica PS: Patients who have undamaged and functional collateral ligaments for the group requiring Physica PS
  Interventions: Device: Physica PS

INTERVENTIONS:
Device: Physica CR — Cruciate retaining total knee replacement
  Groups: Physica CR
Device: Physica PS — Posterior Stabilized total knee replacement
  Groups: Physica PS

SUMMARY:
Type & Design:

Post-market, international, multicentre Prospective, parallel groups, open-label, baseline controlled

Objectives:

1. Assessment of clinical, radiographic and patient-reported outcomes of Physica CR and PS designs
2. Incidence of adverse events and identification of possible risk factors for unsatisfactory results
3. Mid-term survivorship of the implants

ELIGIBILITY:
Inclusion Criteria:

1. Male and females
2. Age 22-78 years
3. Any race
4. Ambulatory patients
5. Patients who have a medical condition with over 5 years of life expectancy
6. Patients with painful primary or secondary knee osteoarthritis
7. Patients who have undamaged and functional collateral and posterior cruciate ligaments for the group requiring Physica CR or Patients who have undamaged and functional collateral ligaments for the group requiring Physica PS
8. Patients with flexion ≥90° on the affected side
9. Patients with a fixed flexion contracture <20°
10. Patients who understand the conditions of the study and are willing and able to comply with the prescribed rehabilitation and to perform all scheduled follow-up visits
11. Patients who have signed the Ethics Committee approved study-specific Informed Consent Form prior to the surgery

Exclusion Criteria:

1. Previous partial knee replacement or patellofemoral joint replacement and previous patellectomy
2. Primary Total Knee Replacement (TKR) in the affected knee
3. Varus deformity >20° or Valgus deformity >15°
4. Patients with a fixed flexion contracture >20°
5. Previous intra-articular fractures of the affected knee
6. Patients with previous methaphysal tibial or femoral osteotomy performed less than 5 years before the screening visit, in case of plate removal surgery it is done early than 1 year ago to screening.
7. Previous knee replacement on the contralateral side within the last year and whose outcome is achieving an KSS< 60 points
8. Patients with symptomatic Osteoarthritis (OA) of the spine if the assessment of pain with Numeric Rating Scale is >4
9. Patients with an history of infections (on the affected knee or systemic)
10. Muscular insufficiency or absence of muscoligamentous supporting structures required for adequate soft tissue balance
11. Patients who have damaged or absence of the posterior cruciate ligament for the group requiring Physica CR
12. Patients with known or suspicious metal hypersensitivity
13. Recurrent medical history of severe allergic or immune-mediated reactions
14. Vascular insufficiency of lower limbs severe enough to interfere with the study evaluation
15. Current treatment or treatment within the previous 2 years before the screening visit for malignant and life-threatening non-malignant disorders
16. Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation including:

    1. any intercurrent chronic disease or condition that may interfere with the completion of the 5-year follow-up, such as liver disease, severe coronary disease, drug or alcohol abuse
    2. significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery
    3. neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
    4. known metabolic disorders leading to progressive bone deterioration
17. Patients who have known co-existent medical condition with less 5 years of life expectancy
18. Previous organ transplant surgery
19. Any psychiatric illness that would prevent comprehension of the details and nature of the study
20. Participation in any experimental drug/device study within the 6 months prior to the screening visit
21. Female patients who are pregnant, nursing, or planning a pregnancy

Ages: 22 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population of subjects requiring a primary TKR with a diagnosis of painful primary or secondary osteoartrithis not responding to other conservative treatments, after the review of medical history and the radiographic evaluation of the affected knee.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical change in Knee Society Score (KSS) | From preoperative (baseline) to 5 years after surgery
  KSS is divided into two components: the first ("Knee Score", KKSS) assesses the knee clinically through the physical examination, and the second ("Function Score", FKSS) assesses the individual's functionality, while both attain a total of 100 points each. The Clinical KSS (KKSS) evaluates pain (50 points), stability (25 points) and range of motion (25 points). The Functional KSS (FKSS) evaluates the walking distance (50 points), and the act of climbing and descending stairs (50 points).
  The system for selecting patients is provided through three categories: A- unilateral or bilateral (opposite knee replaced successfully), B- unilateral, other knee symptomatic and C- polyarthritis or clinical disease.
  Scores rating from 80 to 100 is considered excellent, from 70 to 79 good, from 60 to 69 fair, and less than 60 poor.

SECONDARY OUTCOMES:
Functional change in Timed up and Go (TUG) test | From preoperative (baseline) to 5 years after surgery
  The Timed-get-up-and-go test (TUG) is a simple test widely used to assess a person's mobility, requiring both static and dynamic balance. Subjects are instructed to walk as quickly as they feel safe and comfortable. Time (seconds) is taken to rise from a chair (seat height, 46 cm), walk 3 meters, turn around, walk back to the chair, then sit down wearing regular footwear. The TUG has excellent inter-rater and intra-rater reliability. Timing starts on the signal to start and terminates once the participant sits back down fully with their back resting on the back of the chair. Regular walking aid is allowed and recorded if required. Two trials are performed and the faster of the 2 trials is recorded to nearest 10th of a second.
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) | From preoperative (baseline) to 5 years after surgery
  KOOS was developed and is validated for several cohorts of younger and/or more active patients with knee injury and/or knee osteoarthritis. KOOS is a 42-item self-administered self-explanatory questionnaire that covers five patient-relevant dimensions: Pain, Other Disease-Specific Symptoms, Active Daily Living Function, Sport and Recreation Function, and knee-related Quality of Life. The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures.
Change in Satisfaction Visual Analogue Scale (Satisfaction VAS) | From 3 months to 5 years after surgery
  A Satisfaction Visual Analogue Scale (VAS) system was developed to evaluate patient satisfaction with the TKR at follow-up, similar to the system used to measure pain. The scale consists of a 10-cm-long horizontal line ranging from completely satisfied to totally unsatisfied. On top of the scale the question: "Are you satisfied with your knee prosthesis?" is placed. Facial expressions are put above the line to express satisfaction visually. The patient receives this scale and is asked to mark the line at a point that would match his/her satisfaction. With a ruler, the number of millimetres is measured and converted to points. The satisfaction VAS system ranges from 100 (best, completely satisfied) to 0 (worst, totally unsatisfied) points.
Change in Forgotten Joint Score (FJS-12) | From 3 months to 5 years after surgery
  The Forgotten Joint Scores (FJS-12) comprises measures for the assessment of joint-specific patient-reported outcome and focus on patients' awareness of a specific joint in everyday life. FJS-12 is a 12-item questionnaire that integrates variables such as pain, stiffness, function on activities of daily living, patients' expectations and activity levels and finally psychosocial factors. It consists of 12 questions and is scored using a 5-point Likert response format (never-almost never-seldom-sometimes-mostly) with the raw scores transformed onto a 0-100 point scale. High scores indicate good outcome, that is, a high degree of "forgetting" the joint. FJS-12 evaluation isn't performed preoperatively.
Components stability - radiolucent lines evaluation | From discharge to 5 years after surgery
  The radiographical assessment includes a modified evaluation of presence, location and thickness of periprosthetic radiolucent lines. The sums of the width of radiolucent lines for every component are categorised as follows: 4 or less and non progressive is probably not significant; 5-9 should be closely followed for progression; 10 or greater signifies possible or impending failure regardless of symptoms. Signs of a radiographically loose prosthesis include progressively enlarging luciencies, subsidence of the component or a change in alignment from previous films.
Survival rate of Physica CR and PS | At 3 years and 5 years after surgery
  Survival rate of the implant (Kaplan-Meier)
Incidence of device-related AE/SAE/DD/ADE/SADE | From intraoperative to 5 years after surgery
  Incidence of device-related adverse events( AE), serious adverse events (SAE), device deficiency (DD), adverse device effect (ADE), serious adverse device effect (SADE).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Peretti, MD, Principal Investigator — I.R.C.C.S. Galeazzi (Milan, Italy)
Locations (4):
- Cliniques Universitaires Saint-Luc ASBL, Brussels, Brussels Capital, Belgium
- Italy (2):
  - I.R.C.C.S. Galeazzi, Milan, Milano
  - Casa di cura Citta' di Parma, Parma, Parma
- Clinique d'Eich - centre Hospitalier de Luxembourg, Luxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No